CLINICAL TRIAL: NCT05631262
Title: A Multicenter, Open-label, Phase 2 Study to Evaluate the Efficacy and Safety of SKB264 Monotherapy in Selected Subjects with Advanced Solid Tumors
Brief Title: SKB264 Monotherapy in Selected Subjects with Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅱ-08
Record Dates: First submitted 2022-11-10; First posted 2022-11-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Selected Subjects with Advanced Solid Tumors
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- SKB264 (Cohort 1) (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- SKB264 (Cohort 2) (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- SKB264 (Cohort 3) (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- SKB264 (Cohort 4) (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- SKB264 (Cohort 5) (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- Part II Test group (Experimental): SKB264 will be administered as an intravenous (IV) infusion on Day 1 and Day 15 of each 28-day cycle
  Interventions: Drug: SKB264
- Part II Control group (Active Comparator): Docetaxel will be administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: SKB264 — Subjects of Cohot 1-5 and Part II Test group will receive SKB264 monotherapy
  Arms: Part II Test group; SKB264 (Cohort 1); SKB264 (Cohort 2); SKB264 (Cohort 3); SKB264 (Cohort 4); SKB264 (Cohort 5)
Drug: Docetaxel — Part II Control group will receive docetaxel monotherapy.
  Arms: Part II Control group

SUMMARY:
The purpose of this study is to assess the safety and efficacy of SKB264 monotherapy in subjects with selected advanced solid tumors.The study is divided into two parts: the Part Ⅰ consists of 5 cohorts, and the Part Ⅱ for expansion. Eligible subjects will receive SKB264 monotherapy, until there is no longer clinical benefit, intolerable toxicity, discontinuation of study treatment required by the subject, or other protocol-specified treatment discontinuation criteria, whichever occurs first.

DETAILED DESCRIPTION:
The second part of this study is a randomized, open-label, multicenter Phase 2 clinical study of SKB264 monotherapy versus docetaxel in subjects with locally advanced or metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 to ≤ 75 years at the time of signing the ICF;
2. The following histologically or cytologically confirmed tumor types will be enrolled:

   * Part Ⅰ Cohort 1, Cohort 2, Cohort 3, Cohort 5 and Part Ⅱ: histologically or cytologically confirmed Non Small Cell Lung Cancer (NSCLC);
   * Part Ⅰ Cohort 4: histologically or cytologically confirmed nonkeratinizing differentiated or undifferentiated nasopharyngeal carcinoma (NPC) ;
3. For subjects enrolled in Part I Cohort 1 and Part II, the following criteria must be met:①EGFR-sensitive mutations confirmed by tumor histology or cytology or hematology;②Failure of prior EGFR-TKI therapy and chemotherapy;
4. For subjects enrolled in Part I Cohort 2, the following criteria must be met:①EGFR-sensitive mutations confirmed by tumor histology or cytology or hematology;②Failure of prior EGFR-TKI therapy;③No prior systemic therapy for locally advanced or metastatic NSCLC other than EGFR-TKI therapy;
5. For subjects enrolled in Part I Cohort 3, the following criteria must be met:

   ①NSCLC confirmed by tumor histology to be EGFR wild-type and negative for ALK fusion gene; ②Subjects must have met one of the following conditions for prior systemic therapy:A. Have received platinum-based chemotherapy in combination with anti-PD-1/L1 monoclonal antibody therapy as the only prior first-line therapy;B. Have received sequential treatment with platinum-based chemotherapy and anti-PD-1/L1 monoclonal antibody (in either order) as the only prior second-line therapy;
6. For subjects enrolled in Part I Cohort 4, the following criteria must be met:

   Have received prior second-line or above systemic therapies and have progressed on or after treatment, with prior therapies including platinum-based chemotherapy and anti-PD-1/PD-L1 monoclonal antibody therapy;
7. For subjects enrolled in Part I Cohort 5, the following criteria must be met:

   ①The presence of other driver gene alterations confirmed by tumor histology or cytology or hematology other than EGFR-sensitive mutations ;②have failed targeted therapy for applicable genetic alterations or chemotherapy;
8. PD as assessed by imaging on or after the most recent treatment for locally advanced or metastatic disease;
9. Ability to provide fresh or archival tumor tissue for biomarker testing and analysis.
10. At least one measurable target lesion per RECIST 1.1;
11. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
12. Expected survival ≥ 12 weeks;
13. Adequate organ and bone marrow function;
14. Female subjects of childbearing potential and male subjects with partners of childbearing potential who use effective medical contraception during the study treatment period and for 6 months after the end of dosing;
15. Subjects who voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol- specified visits and relevant procedures.

Exclusion Criteria:

1. For NSCLC, histologically or cytologically confirmed the presence of small cell lung cancer, neuroendocrine carcinoma, and carcinosarcoma components;
2. Subjects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression, or active brain metastases.
3. Other malignancies within 3 years prior to the first dose;
4. Presence of any cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors:
5. Uncontrolled systemic disease as judged by the investigator:
6. History of (noninfectious) interstitial pneumonia (ILD)/noninfectious pneumonitis requiring steroid therapy and current ILD/noninfectious pneumonitis, or suspected ILD/noninfectious pneumonitis at screening that cannot be excluded by imaging;
7. Clinically serious lung injuries caused by lung diseases, including but not limited to any underlying lung diseases or prior pneumonectomy;
8. Presence of active chronic inflammatory bowel disease, GI tract obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute GI tract bleed;
9. Toxicities treated by prior anti-tumor therapy having not recovered to ≤ Grade 1 (as per NCI CTCAE V5.0) or to the levels specified in the eligibility criteria;
10. Presence of active hepatitis B or hepatitis C;
11. Subjects with HIV test positive or history of AIDS; known active syphilis infection;
12. Known allergy to the study drug or any of its components, and a history of known severe hypersensitivity to other monoclonal antibodies;
13. Prior TROP2-targeted therapy;
14. Prior treatment with any drug therapy targeting topoisomerase I inhibitor, including antibody-drug conjugates (ADCs);
15. Major surgery within 4 weeks prior to the first dose or expected to require major surgery during the study;
16. Systemic anti-infective therapy within 2 weeks prior to the first dose;
17. Receipt of any systemic anti-tumor therapy such as macromolecular targeted therapy, immunotherapy, etc. within 4 weeks prior to the first dose; receipt of small molecule TKIs, nonspecific immunomodulatory therapy , and Chinese patent drug preparations for approved anti-tumor indications within 2 weeks prior to the first dose;
18. Ongoing long-term systemic corticosteroid therapy of > 10 mg prednisone or equivalent dose of systemic corticosteroids or equivalent anti-inflammatory active medication or any form of immunosuppressive therapy prior to the first dose;
19. Live vaccines inoculated within 30 days prior to the first dose or planned to be inoculated during the study;
20. Rapid deterioration of disease, such as significant changes in performance status during the screening process prior to the first dose;
21. Pregnant or lactating women;
22. Presence of local or systemic diseases caused by non-malignancies; or diseases or symptoms secondary to tumors that can lead to high medical risks and/or uncertainties in survival evaluation;
23. Any condition that, in the opinion of the investigator, make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 21 months.
  ORR is defined as the proportion of subjects with confirmed complete response (CR) or partial response (PR) as the best overall response assessed per RECIST 1.1.
Incidence and severity of adverse events (AEs) | From subject sign the informed consent form (ICF) to 30 days after the last dose of study treatment.
  Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From baseline until disease progression, death, or other protocol defined reason,up to approximately 21 months.
  PFS is defined as the time from the first dose to progressive disease (PD) or death, whichever occurs first. PD will be assessed per RECIST 1.1.
Duration of response (DOR) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 21 months.
  DOR is defined as the time from the date of first documented CR or PR to PD or death due to any cause, whichever occurs first.
Disease control rate (DCR) | From baseline until disease progression, death, or other protocol defined reason, up to approximately 21 months.
  DCR is defined as the proportion of subjects with CR, PR or stable disease (SD) as the best overall response assessed per RECIST 1.1.
Overall survival (OS) | From baseline until death due to any cause.
  OS is defined as the time period from the start of administration to death due to any cause.
Immunogenicity | From baseline up to 12 months after last patient enrollment.
  Presence of Anti-drug antibodys (ADAs) for SKB264.
PK | From baseline up to 12 months after last patient enrollment.
  Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) of SKB264-ADC, SKB264-TAB and free KL610023.
PK | From baseline up to 12 months after last patient enrollment.
  Pharmacokinetic Parameter Minimum Plasma Concentration (Cmin) of SKB264-ADC, SKB264-TAB and free KL610023.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Fang W, Li X, Wang Q, Meng X, Zheng W, Sun L, Yao W, Zhuang W, Fan Y, Zhuo M, Luo Y, Zhang Z, Song X, Yang R, Yang J, Jin X, Diao Y, Ge J, Zhang L. Sacituzumab tirumotecan versus docetaxel for previously treated EGFR-mutated advanced non-small cell lung cancer: multicentre, open label, randomised controlled trial. BMJ. 2025 Jun 5;389:e085680. doi: 10.1136/bmj-2025-085680. PMID 40473437
- [Derived] Zhao S, Cheng Y, Wang Q, Li X, Liao J, Rodon J, Meng X, Luo Y, Chen Z, Wang W, Yi T, Li Y, Yin Y, Xu H, Yu G, Mi Y, Fan Y, Wainberg ZA, Wang X, Su C, Yu Q, Lai S, Sun L, Zhuang W, Wang X, Yang J, Li Y, Ge J, Li J, Zhang L, Fang W. Sacituzumab tirumotecan in advanced non-small-cell lung cancer with or without EGFR mutations: phase 1/2 and phase 2 trials. Nat Med. 2025 Jun;31(6):1976-1986. doi: 10.1038/s41591-025-03638-2. Epub 2025 Apr 10. PMID 40210967